CLINICAL TRIAL: NCT01055535
Title: An Open Label, Single Centre Trial of Microplasmin Intravitreal Injection for Non-Surgical Treatment of Focal Vitreomacular Adhesion
Brief Title: Safety and Efficacy Study of Microplasmin in for Non-Surgical Treatment of Focal Vitreomacular Adhesion
Acronym: MIVI-8
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-MV-008
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Focal Vitreomacular Adhesion
MeSH Terms: interventions — microplasmin

ARMS (1):
- Microplasmin (Experimental)
  Interventions: Drug: Microplasmin

INTERVENTIONS:
Drug: Microplasmin — 125 µg intravitreal injection

SUMMARY:
This study will evaluate the safety and efficacy of Microplasmin administered as an intravitreal injection, in subjects with focal vitreomacular adhesion. Ultimately, it is believed that intravitreal microplasmin may offer physicians a safe agent for pharmacologic vitreolysis and induction of Posterior Vitreous Detachment (PVD) without the need for vitrectomy. This clinical study is justified because the study sponsor believes the potential benefits outweigh the potential risks, as outlined below.

ELIGIBILITY:
Inclusion Criteria:

* I. Male or female patients aged > 18
* II. Presence of focal vitreomacular adhesion (ie, central vitreal adhesion within 6mm OCT field surrounded by elevation of the posterior vitreous cortex
* III. BCVA of 20/32 or worse in the study eye
* IV. BCVA of 20/400 or better in the contralateral eye
* V. Written informed consent obtained from the patient prior to inclusion in the study

Exclusion Criteria:

* I. Evidence of complete macular PVD in the study eye on biomicroscopy, B-scan or OCT prior to planned study drug injection
* II. Any evidence of proliferative retinopathy meeting the definition for PDR in the study eye
* III. Patients with vitreous hemorrhage which precludes either of the following: visualization of the posterior pole by visual inspection OR adequate assessment of the macula by either OCT and/or fluorescein angiogram in the study eye
* IV. Patients with rhegmatogenous retinal detachment, PVR, or retinal degenerative changes associated with increased risk of retinal detachment in the study eye. Such retinal degenerative changes include lattice degeneration or cystic retinal tufts. Thorough retinal examination should be performed in all patients to rule out these changes.
* V. Patients with high myopia (> 8D) or aphakia in the study eye

VI. Patients with history of rhegmatogenous retinal detachment in the fellow eye VII. Patients who have had ocular surgery in the study eye in the prior three months VIII. Patients who have had a vitrectomy in the study eye at any time. IX. Patients with glaucoma that is not controlled with topical medication or that is associated with severe visual field loss, documented by perimetry, in the study eye X. Patients who have had laser photocoagulation treatment in the study eye in the previous 3 months XI. Intravitreal injection of any drug in the study eye in the previous 3 months XII. Patients who are pregnant or of child-bearing potential not utilizing a form of contraception acceptable to the Investigator XIII. Patients who, in the investigators view, will not complete all visits and investigations, including the last visit at 6 months after the last injection XIV. Patients who have participated in an investigational drug study within the past 30 days XV. Patients with hypertension (either SBP > 170 or DBP > 100 mm Hg) XVI. Patients with a life expectancy less than 6 months XVII. Patients who have previously participated in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
History/full ophthalmologic examination (including full retinal examination: baseline, post-injection days 7, 14 and 28 and months 3 and 6 | baseline, day 7, 14 and 28 and months 3 and 6

SECONDARY OUTCOMES:
Proportion of patients with nonsurgical resolution of focal vitreomacular adhesion at study visits other than the 28 day post-injection visit | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium